CLINICAL TRIAL: NCT00003992
Title: Pilot Trial of Paclitaxel-Herceptin Adjuvant Therapy for Early Stage Breast Cancer
Brief Title: Chemotherapy Plus Monoclonal Antibody Therapy in Treating Women With Stage II or Stage IIIA Breast Cancer That Overexpresses HER2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02305; E-2198; CDR0000067197 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Cyclophosphamide; Doxorubicin; Paclitaxel; Tamoxifen

ARMS (2):
- Arm I (Experimental): Patients receive paclitaxel IV over 3 hours immediately followed by trastuzumab (Herceptin) IV over 30-90 minutes on day 1. Paclitaxel repeats every 3 weeks for 4 courses and trastuzumab (Herceptin) repeats weekly for 10 courses. At 3 weeks following paclitaxel and trastuzumab (Herceptin), patients receive doxorubicin IV and cyclophosphamide IV over 1 hour every 3 weeks for 4 courses. Following chemotherapy, estrogen receptor (ER) positive and/or progesterone receptor (PR) positive patients receive oral tamoxifen twice daily for 5 years.
  Interventions: Biological: trastuzumab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel; Drug: tamoxifen citrate
- Arm II (Experimental): Patients receive same therapy as in Arm I, except for additional trastuzumab (Herceptin) IV weekly beginning within 3 weeks following completion of chemotherapy and local therapy and continuing for 1 year. ER and/or PR positive patients receive tamoxifen as in Arm I but may be concurrent with trastuzumab (Herceptin). Following completion of doxorubicin and cyclophosphamide, post lumpectomy and post mastectomy patients may receive local radiotherapy daily for 5-6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Biological: trastuzumab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: paclitaxel
Drug: tamoxifen citrate
  Arms: Arm I

SUMMARY:
Randomized phase II trial to study the effectiveness of chemotherapy with paclitaxel and the monoclonal antibody trastuzumab followed by chemotherapy in treating women who have stage II or stage IIIA breast cancer that overexpresses HER2. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies can locate tumor cells and deliver tumor-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the safety of paclitaxel plus trastuzumab (Herceptin) followed by adjuvant chemotherapy in women with node positive stage II or IIIa breast cancer with HER2 overexpression.

II. Evaluate the safety of long term trastuzumab (Herceptin) in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to radiotherapy (none planned vs planned to breast or chest wall). Patients are randomized to one of two treatment arms.

ARM I: Patients receive paclitaxel IV over 3 hours immediately followed by trastuzumab (Herceptin) IV over 30-90 minutes on day 1. Paclitaxel repeats every 3 weeks for 4 courses and trastuzumab (Herceptin) repeats weekly for 10 courses. At 3 weeks following paclitaxel and trastuzumab (Herceptin), patients receive doxorubicin IV and cyclophosphamide IV over 1 hour every 3 weeks for 4 courses. Following chemotherapy, estrogen receptor (ER) positive and/or progesterone receptor (PR) positive patients receive oral tamoxifen twice daily for 5 years.

ARM II: Patients receive same therapy as in Arm I, except for additional trastuzumab (Herceptin) IV weekly beginning within 3 weeks following completion of chemotherapy and local therapy and continuing for 1 year. ER and/or PR positive patients receive tamoxifen as in Arm I but may be concurrent with trastuzumab (Herceptin). Following completion of doxorubicin and cyclophosphamide, post lumpectomy and post mastectomy patients may receive local radiotherapy daily for 5-6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 200 patients (100 per treatment arm) will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II or IIIa (T1-T3, N1-N2, M0) adenocarcinoma of the breast HER2 overexpression (2-3+ by immunochemistry)
* Bilateral breast cancer allowed
* Must have had local breast cancer surgery within past 12 weeks
* Mastectomy or lumpectomy with clear surgical margins AND axillary lymph node dissection with at least 6 nodes removed
* Hormone receptor status: Not specified

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Sex: Female
* WBC at least 3,000/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9 g/dL
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Creatinine no greater than 1.5 times ULN
* LVEF at least 50%
* No history of congestive cardiomyopathy
* No congestive heart failure or myocardial infarction within the past 6 months
* No uncontrolled hypertension
* No uncontrolled arrhythmia within the past 6 months
* No other prior malignancy within the past 5 years except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No other serious medical illness that would limit survival to less than 2 years
* No psychiatric condition precluding study
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for breast cancer
* No prior hormonal therapy for breast cancer
* At least one year since prior tamoxifen for chemoprevention (e.g., Breast Cancer Prevention Trial)
* No prior radiotherapy to the breast, chest wall, or regional lymph nodes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 1999-08; Primary Completion 2007-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George W. Sledge, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (45):
- United States (44):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Hunterdon Regional Cancer Program, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - Kaplan Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Sledge GW, O'Neill A, Thor A, et al.: Adjuvant trastuzumab: long-term results of E2198. [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-2075, S106, 2006.